CLINICAL TRIAL: NCT06068946
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, 13-week Study of VK2735 for Weight Management in Subjects Who Are Obese, or Overweight With at Least One Weight-related Comorbid Condition
Brief Title: VK2735 for Weight Management Phase 2
Acronym: VENTURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VK2735-201
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Weight Loss
Keywords: Overweight; Obese
MeSH Terms: conditions — Weight Loss; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VK2735 (Placebo) (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- VK2735 (Dose #1) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist
  Interventions: Biological: VK2735
- VK2735 (Dose #2) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist
  Interventions: Biological: VK2735
- VK2735 (Dose #3) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist
  Interventions: Biological: VK2735
- VK2735 (Dose #4) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist
  Interventions: Biological: VK2735

INTERVENTIONS:
Biological: VK2735 — VK2735 is a peptide GLP-1 and GIP dual agonist
  Arms: VK2735 (Dose #1); VK2735 (Dose #2); VK2735 (Dose #3); VK2735 (Dose #4)
Biological: Placebo — Placebo comparator
  Arms: VK2735 (Placebo)

SUMMARY:
This is a phase 2, 13-week randomized, double-blind, placebo-controlled, parallel arm study that will evaluate the safety, tolerability, weight loss efficacy, pharmacodynamic effects, and pharmacokinetics of VK2735 in adults who are obese (BMI ≥30 kg/m2) or who are overweight (BMI ≥27 kg/m2) with at least one weight-related co-morbid condition.

VK2735 or matched placebo will be administered once weekly.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of signing the informed consent
2. Body mass index (BMI) ≥30 kg/m2 OR ≥27 kg/m2 with at least one weight-related co-morbid condition (treated or untreated), and BMI <50 kg/m2

Exclusion Criteria:

1. History of or current clinically significant medical or psychiatric disorder that, in the opinion of the Investigator, does not support study participation
2. Self-reported body weight change of 5% or more within 3 months of screening
3. Current or past diagnosis of diabetes mellitus (including type 1, type 2, gestational)
4. Current or past diagnosis of chronic pancreatitis
5. Calcitonin ≥20 ng/L measured by central laboratory at screening (individuals with elevated calcitonin at initial screening may be re-screened)
6. Any GLP-1 receptor agonist or GLP-1/GIP dual agonist within 6 months of Screening
7. Any prescription or over-the-counter medications intended for weight loss within 6 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Percent (relative) change from baseline to Week 13 in body weight | 13 weeks
  To measure the efficacy of VK2735 for weight loss in adult Subjects who are obese, or overweight with at least one weight-related comorbid condition

SECONDARY OUTCOMES:
Proportion of Subjects losing ≥5% and ≥10% of baseline weight at Week 13 | 13 weeks
  To measure the efficacy of VK2735 for weight loss in adult Subjects who are obese, or overweight with at least one weight-related comorbid condition

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), TESAEs, AESI | 13 weeks
  To evaluate the safety and tolerability of VK2735 for weight loss in adult Subjects who are obese, or overweight with at least one weight-related comorbid condition

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Viking Clinical Site #119, Birmingham, Alabama
  - Viking Clinical Site #114, Long Beach, California
  - Viking Clinical Site #110, Los Angeles, California
  - Viking Clinical Site #113, Tustin, California
  - Viking Clinical Site #116, Clearwater, Florida
  - Viking Clinical Site #106, Clearwater, Florida
  - Viking Clinical Site #112, Jacksonville, Florida
  - Viking Clinical Site #105, Ocoee, Florida
  - Viking Clinical Site #107, Port Orange, Florida
  - Viking Clinical Site #104, Indianapolis, Indiana
  - Viking Clinical Site #103, Louisville, Kentucky
  - Viking Clinical Site #109, Marrero, Louisiana
  - Viking Clinical Site #102, Kansas City, Missouri
  - Viking Clinical Site #111, Butte, Montana
  - Viking Clinical Site #108, Knoxville, Tennessee
  - Viking Clinical Site #101, Austin, Texas
  - Viking Clinical Site #118, Austin, Texas
  - Viking Clinical Site #100, Phoenix, Texas
  - Viking Clinical Site #115, San Antonio, Texas
  - Viking Clinical Site #117, San Antonio, Texas

REFERENCES:
- [Derived] Bays HE, Toth P, Alkhouri N, Pullman J, Freilich B, Neutel J, Ji S, Stubbe S, Hedges P, Lian B. Weekly Subcutaneous VK2735, a GIP/GLP-1 Receptor Dual Agonist, for Weight Management: Phase 2, Randomized, 13-Week VENTURE Study. Obesity (Silver Spring). 2026 Jan 8. doi: 10.1002/oby.70106. Online ahead of print. PMID 41508550